CLINICAL TRIAL: NCT06980727
Title: Increment Value of Intravenous Dexametasone Versus Nebulized Salbutamol for Renal Colic Pain Management in the Emergency Department: A Randomized Clinical Trial
Brief Title: Comparative Efficacy of IV Dexamethasone vs. Nebulized Salbutamol for Renal Colic Pain in the ED
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Professor, University of Monastir
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: Renal Colic Salbutamol
Record Dates: First submitted 2025-05-07; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Renal Colic
Keywords: Renal Colic; Salbutamol; Dexamethasone
MeSH Terms: conditions — Renal Colic | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo group (Placebo Comparator): In this group patient will receive 1000mg intravenous injection of paracetamol in combination with 4ml intravenous normal saline as placebo, and 5ml nebulisation of normal saline during 10min.
  Interventions: Drug: Placebo
- Dexamethasone group (Active Comparator): In this group, patients will receive 1000mg intravenous injection of paracetamol in combination with 4ml intravenous dexamethasone (8mg), and 5ml nebulisation of of normal saline during 10min as placebo.
  Interventions: Drug: Dexamethasone
- Salbutamol group (Active Comparator): In this group, patients will receive 1000mg intravenous injection of paracetamol in combination with 4ml IV normal saline as placebo, and 5mg salbutamol in 5ml nebulisation during 10min
  Interventions: Drug: Salbutamol 2,5 mg

INTERVENTIONS:
Drug: Salbutamol 2,5 mg — In this study group, patients will receive 1000mg intravenous injection of paracetamol in combination with 4ml IV normal saline as placebo, and 5mg salbutamol in 5ml nebulisation during 10min.
  Arms: Salbutamol group
Drug: Dexamethasone — Patients will receive 1000mg intravenous injection of paracetamol in combination with 4ml intravenous dexamethasone (8mg), and 5ml nebulisation of of normal saline during 10min as placebo.
  Arms: Dexamethasone group
Drug: Placebo — Patients will receive 1000mg intravenous injection of paracetamol in combination with 4ml intravenous dexamethasone (8mg), and 5ml nebulisation of of normal saline during 10min as placebo.
  Arms: Placebo group

SUMMARY:
Adult patients (18-55 years of age) with clinical diagnosis of acute renal colic (sudden sharp colic flank pain with or without radiation to genitalia or groin and with or without urinary symptoms) who had pain score of 5 or more measured by 10-cm visual analogue scale (VAS), will be included. Will be excluded those who had history of cardiovascular, hepatic, renal or metabolic diseases, patients with evidence of sepsis or clinical suspicion of urinary tract infection, hemodynamically unstable patients (systolic blood pressure <90 mmHg), patients with uncontrolled diabetes, pregnancy, breastfeeding, patients unable to understand verbal and/or written information, patients receiving analgesics within 6 hours before presentation, serum potassium less than 3.7 mmol/l, concomitant use of any beta blockers (including beta-blocker containing eye drops), prolonged-release long-acting β-agonists, use of short-acting β2-agonists within the 6 h preceding presentation to the emergency department, any contraindication to the use of salbutamol, history of drug dependence or chronic consumption of alcohol. Will be also excluded patients with known allergy to paracetamol or salbutamol, patients with abdominal tenderness as a sign of peritoneal inflammation and those with any clinical suspicion for diseases other than urolithiasis, including abdominal aortic aneurysm or dissection.

ELIGIBILITY:
Inclusion criteria:

* Adults aged 18-65 years
* Clinical diagnosis of acute renal colic (defined as sudden sharp colicky flank pain with or without radiation to the genitalia or groin, and with or without urinary symptoms)
* Pain score of 5 or more measured using the 10-cm NRS scale

Exclusion Criteria:

* History of cardiovascular, hepatic, renal, or metabolic diseases
* Evidence of sepsis or clinical suspicion of urinary tract infection
* Hemodynamically unstable (systolic blood pressure < 90 mmHg)
* Uncontrolled diabetes
* Pregnancy or breastfeeding
* Inability to understand verbal and/or written information
* Received any analgesics within 6 hours prior to presentation
* Serum potassium < 3.7 mmol/L
* Concomitant use of:

Any beta-blockers (including beta-blocker-containing eye drops)

Prolonged-release long-acting β-agonists

Short-acting β2-agonists within 6 hours prior to presentation

* Contraindication to salbutamol use
* Known allergy to paracetamol or salbutamol
* Abdominal tenderness suggestive of peritoneal inflammation
* Clinical suspicion of conditions other than urolithiasis, including:
* Abdominal aortic aneurysm
* Aortic dissection
* History of drug dependence or chronic alcohol consumption

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Change level of NRS by 50%. | 120 minutes post-intervention
  The efficacy of the drug with regards to reducing the Numerical Rating Scale (NRS) A scale from 0 to 10 with 0 meaning "no pain" and 10 meaning "worst imaginable pain."during the follow-up. Criteria for treatment response was determined as pain reduction level by 50% based on the primary NRS score or NRS score of four or lower.

SECONDARY OUTCOMES:
Adverse effects | 120 minutes post-intervention
  The occurrence of adverse effects
Rescue analgesia. | 120 minutes post-intervention
  The number of patients who need rescue analgesia.